CLINICAL TRIAL: NCT04404738
Title: Clinical Studies of Robotic-assisted Surgery in Urology With MicroPort® Endoscopic Instrument Control System
Brief Title: MicroPort® Endoscopic Instrument Control System to Accomplish Robotic-assisted Surgery in Urology
Acronym: MARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Gao Xu, Chief Physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPMB-2019-MKW
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Robotic Surgical Procedures; Prostatectomy; Nephrectomy
Keywords: robot; efficacy; safety; urology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MicroPort® Surgical System (Experimental): robot-assisted surgeries, for instance, prostatectomy, cystectomy or nephrectomy will be performed using MicroPort® surgical system
  Interventions: Procedure: MicroPort® robot-assisted laparoscopic surgery
- da Vinci Surgical System (Active Comparator): robot-assisted surgeries, for instance, prostatectomy, cystectomy or nephrectomy will be performed using da Vinci surgical system
  Interventions: Procedure: da Vinci robot-assisted laparoscopic surgery

INTERVENTIONS:
Procedure: MicroPort® robot-assisted laparoscopic surgery — In this group, patients undergoing robot-assisted laparoscopic surgery in urology will be performed by Microport® Surgical System
  Arms: MicroPort® Surgical System
Procedure: da Vinci robot-assisted laparoscopic surgery — In this group, patients undergoing robot-assisted laparoscopic surgery in urology will be performed by da Vinci Surgical System
  Arms: da Vinci Surgical System

SUMMARY:
Laparoscopy, now virtually completely, was replaced with robotic surgery in uro-oncological surgery in the world. And given the significant increase in the number of robotic surgeries for prostate, bladder and kidney cancer, it is now a major domain in oncological surgery. Microport MedBot Inc. has independently developed a domestic surgical robot in China. Therefore, the purpose of the study is to evaluate the safety and efficacy of the Chinese robot when applied to surgery in oncology.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 18 years and 80 years;
* laparoscopic surgery is required with one of the following surgical indications:(1)planning to perform radical prostatectomy(clinical stage is T1 or T2,and PSA≥ 0.2ng/mL) ;(2) planning to perform nephrectomy
* being able to cooperate and complete the follow-up and related examinations;
* volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

* patients requiring emergency surgery;
* have severe cardiovascular or circulatory disease and cannot tolerate surgery;
* participated in other clinical trials in the last 3 months;
* failure to understand study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
surgical success rate | 24 hours following the surgery
  Surgery is completed without conversion to other operations and without a re-operation caused by intraoperative complications within 24 hours

SECONDARY OUTCOMES:
blood loss | during the surgery
  Amount of intraoperative bleeding in the patient from the start to the end of the operation
operative time | during the surgery
  The starting point and end point of the operation time are the first effective movement of the robot arm and the movement stop of the robot arm after the operation.
length of hospital stay | 24 hours after discharge
  The total hospital days of subjects from the day of the operation to discharge.
perioperative complication rate | 2 weeks after operation
  The overall incidence of intraoperative and postoperative complications.
The physiological load of the surgeon during the surgery | immediately after the surgery
  The physiological load is assessed by the LED scale immediately after the surgery. LED is the local experienced discomfort scale used to assess the intraoperative physiological load of different parts of the surgeon's body. There are 10 points in the scale, and higher score means worse, with 0 means no discomfort and 10 is the worst discomfort.
The psychological load of the surgeon during the surgery | immediately after the surgery
  The psychological load is assessed by the SME scale immediately after the operation. SME scale is the subjective mental effort scale used to assess the intraoperative psychological load of the surgeon. The scale has a total of 150 points, with a scale of 10 points. The higher the score, the worse it is, with 0 means no any difficult and above 110 points means extremely difficult.
the critical failure rate of the robotic system | during the surgery
  Critical failures that are difficult to repair in a short period of time during robot-assisted surgery and can have a serious impact on the process or the operation
the recoverable malfunction rate of the robotic system | during the surgery
  Recoverable malfunction meant minor errors that could be easily resolved by the technician and has no significant impact on the process or the operation
Instrument performance | immediately after the surgery
  The researcher fills in the instrument performance evaluation form after the operation to review the performance of the instrument during the test.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Gao, professor, Principal Investigator — Changhai Hospital; Jianming Guo, professor, Principal Investigator — Shanghai Zhongshan Hospital; Wei Xue, professor, Principal Investigator — RenJi Hospital
Locations (4):
- China (4):
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - The first affiliated hospital of naval medical university (Shanghai changhai hospital), Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Zhejiang Provincial People's Hospital, Zhejiang

IPD SHARING:
Plan to Share IPD: No